CLINICAL TRIAL: NCT05928897
Title: Efficacy and Safety of Disitamab Vedotin Combined With Sintilimab in Second-line Treatment of Advanced Gastric Cancer: a Prospective, Single Arm Clinical Study (DVES)
Brief Title: Efficacy and Safety of Disitamab Vedotin Combined With Sintilimab
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, zlkzengshan, Director, Xiangya Hospital of Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202208181
Record Dates: First submitted 2023-06-25; First posted 2023-07-03 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer, Her-2, ADC
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamab Vedotin Combined With Sintilimab (Experimental): Disitamab Vedotin (2.5mg/kg, ivgtt, Q3W) Combined With Sintilimab (200mg, ivgtt, Q3W) untill diseases progress
  Interventions: Drug: Disitamab Vedotin combined with Sintilimab

INTERVENTIONS:
Drug: Disitamab Vedotin combined with Sintilimab — Disitamab Vedotin combined with Sintilimab
  Other Names: RC48

SUMMARY:
Efficacy and Safety of Disitamab Vedotin Combined With Sintilimab in Second-line Treatment of Advanced Gastric Cancer: a Prospective, Single Arm Clinical Study

DETAILED DESCRIPTION:
We initiated the efficacy and safety of the first Disitamab Vedotin combined with Sintilimab in second-line therapy in patients with advanced gastric cancer with positive HER2 or low expression of HER2.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric adenocarcinoma, which is diagnosed as unresectable locally advanced, recurrent or metastatic gastric and gastroesophageal junction adenocarcinoma (including signet-ring cell carcinoma, mucinous adenocarcinoma, hepatoid adenocarcinoma).
* Pathological results showed that the expression of HER-2 was positive (IHC score 3+, or IHC score 2+ and ISH score positive) or low (IHC score 1+, or IHC score 2+ and ISH score negative) in gastric adenocarcinoma.
* Failed to receive first-line system medication of gastric carcinoma chemotherapy.
* Male or female, aged 18-75 years old.
* ECOG score 0-2.
* Life expectancy more than 12 weeks.
* There is at least one measurable or assessable focus (According to RECIST 1.1).
* Patients who received radical radiotherapy within 3 months before entering the study are eligible to participate in this study if the radiation area of bone marrow is less than 30%.
* The function of main organs and bone marrow function are normal, defined as follows:
* Blood test:

  * White blood cell (WBC) ≥ 4.5*103 / mm3;
  * Absolute neutrophil count (ANC) ≥ 1.5*103 / mm3;
  * Blood platelet count ≥ 100*103 / mm3;
  * hemoglobin ≥ 9.0g/dL (no transfusion or erythropoietin dependence within 7 days).
* Liver function:

  * Serum total bilirubin (TBIL) ≤ 1.5 times of upper limit of normal (ULN);
  * Serum Aspartate Transaminase (AST) and serum Alanine Aminotransferase For patients without liver metastasis, Transaminase (ALT) ≤ 2.5 times of ULN;
  * For patients with liver metastasis, ALT or AST ≤ 5 times of ULN.
* Renal function:

  * Serum creatinine (Cr) ≤ 1.5 times of ULN or Cr clearance ≥ 60 mL/min (Cockcroft-Gault formula);
  * Urinary protein (UPRO) < 2+ or Quantification of 24-hour urinary protein < 1g.
* Coagulation function:

  * International normalized ratio (INR) ≤ 1.5 times of ULN or prothrombin time (PT) ≤ 1.5 times of ULN; within 7 days before treatment.
  * If the subject is receiving anticoagulant therapy, PT is within the range of anticoagulant.
* Cardiac function:

  * New York Heart Association (NYHA) grade < 3;
  * Left ventricular ejection fraction ≥ 50%;
  * The baseline of ECG is no atrioventricular block or PR interval prolongation.
* Pulmonary function:

  * Carbon Monoxide Diffusing Capacity (DLCO) ≥ 70% predicted OR;
  * DLCO < 70% and ≥ 55%, the maximal oxygen consumption (VO2max) ≥ 10 L/min/kg (cardiopulmonary assessment) or 6-minutes walk test over 500 meters;
  * Patients with DLCO under 55% are excluded from this study;
  * Pulse oximetry at walking or rest is over 92%.
* The patient and her/his mate should agree to contracept for the time of the study period and within six months after the study (see Section 4.3).
* Patients join the study voluntarily, sign the informed consent file, and be able to comply with the visit and related procedures stipulated in the program.

Exclusion criteria:

* Signs of active bleeding in the focus.
* Previously received anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody, anti-CD137 antibody, anti-CTLA-4 antibody, or other antibodies or drugs targeting T cell costimulatory or checkpoint pathways.
* Be allergic to the active ingredients or excipients of Sintilimab or disitamab vedotin;
* Participate in another interventional clinical study (except observational clinical study or follow-up phase of an intervention study) at the same time;
* Received systemic treatment with anti-tumor indications of proprietary Chinese medicine or immunomodulatory drugs (eg. thymosin/interferon/interleukin, except drugs used locally to control pleural effusion or ascites) within 2 weeks before the first dose.
* Received immunosuppressive drugs within 4 weeks before the first dose of the study, excluding nasal, inhaled or other topical glucocorticoids or physiological doses of systemic glucocorticoids (i.e., no more than 10mg/d prednisone or equivalent doses of other glucocorticoids), or the use of hormones for the prevention of contrast medium allergy.
* Live attenuated vaccine may be received within 4 weeks before the first dose of study treatment or during the study period.
* Note: inactivated injection virus vaccine for seasonal influenza is allowed.
* Surgical procedures were performed within 4 weeks before the first dose of study treatment, or major surgery was expected during the study treatment;
* Laparoscopic exploratory surgery was performed within 2 weeks before the first dose of study treatment.
* There was toxicity (excluding alopecia, non-clinically significant, and asymptomatic laboratory abnormalities) caused by previous antineoplastic therapy that did not return to Grade 0 or 1 in the NCICTCAEv5.0 before the first dose.
* Patients with symptomatic central nervous system cancer metastasis or cancerous meningitis. For previously treated patients with central nervous system cancer metastasis, if their condition is stable (there is no evidence of imaging progress at least 4 weeks before the first administration of the trial treatment, and repeated imaging tests confirm that there is no evidence of new brain metastasis or enlargement of the original brain metastasis), they can participate in the trial in the case they do not need steroid therapy within 14 days before the first dose of the trial treatment.
* Patients with ascites could be found by physical examination; Only imaging shows a small amount of ascites but no symptoms can be selected.
* Patients with moderate amount of bilateral pleural effusion, or large amount of pleural effusion on one side, or patients who have caused respiratory dysfunction and need drainage.
* Patients with bone metastasis at risk of paraplegia.
* Patients with or suspected autoimmune diseases within 2 years (patients with vitiligo, psoriasis, alopecia or Graves' disease who do not need systematic treatment in the past 2 years, patients with hypothyroidism who only need thyroid hormone replacement therapy and type I diabetes patients who only need insulin replacement therapy can be enrolled in the group).
* History of primary immunodeficiency.
* Active pulmonary tuberculosis.
* History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
* History of human immunodeficiency virus (HIV) infection (i.e. HIV antibody positive).
* Severe infection that is active or poorly controlled clinically.
* Symptomatic congestive heart failure (NYHA grade II-IV) or poorly controlled arrhythmia.
* Arterial hypertension (systolic blood pressure ≥ 160mmHg or diastolic blood pressure ≥ 100mmHg) that is still uncontrolled even with standard treatment.
* Arterial thromboembolism occurred within 6 months, including myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack.
* There is a history of deep venous thrombosis, pulmonary embolism or any other severe thromboembolism within 3 months (implantable venous infusion port or catheter-derived thrombosis, or superficial venous thrombosis is not considered "severe" thromboembolism).
* There are uncontrolled metabolic disorders, other non-malignant organs, systemic diseases or secondary reactions to cancer, which can lead to higher medical risk or uncertainty in survival assessment.
* Hepatic encephalopathy, hepatorenal syndrome, Child-Pugh B grade and higher grade liver cirrhosis.
* History of tumor-related intestinal obstruction (within 3 months before the signing of the informed consent) or the following diseases: inflammatory bowel disease or extensive bowel resection (partial colectomy or extensive small bowel resection, complicated with chronic diarrhea), Crohn's disease, ulcerative colitis.
* Patients with acute or chronic active hepatitis B virus (HBsAg positive and HBVDNA viral load ≥ 200IU/mL or ≥ 103copies / mL) or acute or chronic active hepatitis C virus (HCV antibody positive and HCV RNA positive).
* Active syphilis infections who need treatment.
* There was a history of gastrointestinal perforation or fistula within 6 months before the study, except for surgical resection of the primary focus of gastric cancer.
* Suffering from interstitial lung disease that requires steroid treatment.
* History of other primary malignant tumors, except:
* Complete remission of malignant tumors for at least 2 years before the study and no other treatment was required during the study period
* Non-melanoma skin cancer or malignant freckle-like nevus with adequate treatment and no evidence of disease recurrence.
* Primary cancer with adequate treatment and no evidence of disease recurrence.
* Women who are pregnant or breastfeeding.
* Other acute or chronic diseases, mental disorders or laboratory tests that may lead to drug-related risks or interfere with the interpretation of the results of the study, and patients are classified as ineligible to participate in this study according to the judgment of the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  Objective response rate

SECONDARY OUTCOMES:
PFS | 2 years
  Progression-free survival
OS | 2 years
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Shan Zeng, M.D., Principal Investigator — Xiangya Hospital of Central South University

IPD SHARING:
Plan to Share IPD: No